CLINICAL TRIAL: NCT06519630
Title: REHABOTICS: Integrated Rehabilitation System for People With Motor Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pantelis Syringas (Other)
Collaborators: University of Ioannina (Other); Physioloft, Physiotherapy Center (Unknown); University of Peloponnese (Other); Ostracon Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Pantelis Syringas, Principal Investigator, National Technical University of Athens
Organization: National Technical University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REHABOTICS_2022_01
Record Dates: First submitted 2024-07-09; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Stroke; Spasticity, Muscle; Upper Extremity Dysfunction
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabotics Intervention Group (Experimental): Rehabotics Intervention Group received Physiotherapy through the Rehabotics system.
  Interventions: Device: Rehabotics Physiotherapy
- Traditional Physiotherapy Group (Active Comparator): Traditional Physiotherapy Group received Physiotherapy.
  Interventions: Other: Traditional Physiotherapy

INTERVENTIONS:
Device: Rehabotics Physiotherapy — The intervention will be consisted of sessions for participants in the intervention group which includes a repetition of each of the four Sollerman AR Games named, Wallet, Key, Jar, Screwdriver and one repetition of Balloon Pop. Participants will interact with the AR Box and Block Test (BBT) and the serious games under controlled conditions. A clinician will be present throughout the whole session providing help if participants encounter any difficulties. Following the games, the clinician will initiate a stretching program using the Active Exoskeletal Aid, performing 3 sets of 10 repetitions on the finger flexors of the patient's hand. Each rehabilitation session will last 30 minutes and will be conducted three times a week. Similarly, the traditional physiotherapy training program will be prescribed for the control group and will be consisted of sessions lasting 30 minutes per day, three days per week. Both programs duration will be five weeks.
  Arms: Rehabotics Intervention Group
Other: Traditional Physiotherapy — Similarly, the hand functional training program prescribed for the control group consisted of sessions lasting 30 minutes per day, three days per week. Both programs lasted for five weeks and were designed by two clinical experts.
  Arms: Traditional Physiotherapy Group

SUMMARY:
The goal of the Rehabotics project is the development of a comprehensive rehabilitation system to provide highly individualized treatment of upper limb function in patients with motor disorders due to acquired brain damage (eg stroke) or neurodegenerative disease (eg sclerosis), having as central pillar the integration of robotic systems and support functions. A key part of the proposed system is the development and evaluation of an innovative robotic extraskeletal device that will be applied in the form of a glove to the diseased limb of the neurological patient.

The proposed robotic system:

1. will measure various motor and kinematic parameters of the extremity in order to assess the patient's condition and progress, and
2. will offer a specialized rehabilitation program (therapeutic exercises, retraining of functional movements and support of daily activities) through an interactive virtual environment provided by the Rehabotics platform.

The aim is to provide an environment for the provision of a high level of treatment and support services to patients with hand mobility disorders which will take place both in the clinical environment and in the patient's home through telemedicine applications.

To demonstrate the efficiency of the proposed system, Rehabotics will be applied on post-stoke patients for rehabilitation while also using a control group receiving traditional physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* stroke pathology,
* Ashworth Scale ≤ 3,
* 6 months maximum time since the incident

Exclusion Criteria:

* Presence of neurological pathologies that affect hand motion (Parkinson's disease)
* Musculoskeletal deficits that affect normal finger range of motion (e.g. finger fractures, joint stiffness/pain, arthritis that affect joint motion)
* Ashworth Scale > 3,
* Over 6 months since the incident

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Ashworth Scale measured by physiotherapists | Change from baseline to 5 weeks
  This outcome aims to explore the therapeutic potential of Rehabotics in stroke rehabilitation, demonstrating improved hand motor function through the integration of robotics and Augmented Reality games, measured by Ashworth Scale [AS].
  The AS is a key instrument for evaluating spasticity in individuals with upper extremity mobility challenges during rehabilitation. This assessment uses a scoring system from 0 to 4, where higher scores denote greater difficulty in finger movement, and lower scores indicate easier finger movement.
Box and Block Test score measured by physiotherapists | Change from baseline to 5 weeks
  This outcome aims to explore the therapeutic potential of Rehabotics in stroke rehabilitation, demonstrating improved hand motor function through the integration of robotics and Augmented Reality games, measured by the Box and Block Test [BBT] score.
  The BBT consists of a wooden box divided into two compartments by a partition and includes 150 blocks. During the BBT administration, the patient is instructed to move as many blocks as possible, one by one, from one compartment to the other within 60 seconds. The higher the number of blocks moved indicate better manual dexterity.

SECONDARY OUTCOMES:
Device Evaluation Satisfaction utilizing questionnaires for patients | Administered in the 5th week
  This outcome aims to explore the patient satisfaction with the device. Questionnaires will be utilized to gather detailed feedback from patients. These questionnaires will help capture their experiences, satisfaction, captivation and any challenges encountered during the use of Rehabotics.
  The patient questionnaire will cover:
  Comfort and Usability, Perceived Effectiveness (how patients perceive the impact of Rehabotics in their Rehabilitation progress), Engagement and Motivation, Overall Satisfaction.
  Based on the results obtained from the questionnaires, we will be able to identify potential improvements and enhancements for the device, ensuring it better meets the needs and expectations of patients.
Device Evaluation Satisfaction utilizing questionnaires for physiotherapists | 1 year
  This outcome aims to explore the physiotherapist satisfaction with the device. Questionnaires will be utilized to gather detailed feedback from physiotherapists. These questionnaires will help capture their experiences, satisfaction, captivation and any challenges encountered during the use of Rehabotics.
  The physiotherapist questionnaire will include sections on:
  Ease of Use, Effectiveness, Patient Engagement, Technical Issues, Comparison to Traditional Methods
  The results will help refine the design and functionality of Rehabotics, ultimately contributing to more effective and satisfying rehabilitation tool for clinical use.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Papagiannis, PhD, Principal Investigator — Physioloft
Locations (1):
- Physioloft, Physiotherapy Center, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
Patient data cannot be provided due to confidentiality and privacy regulations designed to protect individuals' personal information. Upon a formal request, data may be able to be provided anonymized to protect patients' privacy.